CLINICAL TRIAL: NCT01523379
Title: Efficiacy of the Selctive COX-2-inhibitor Parecoxibe on the Pathological Low Pressure Pain Threshold (PPT) of Patients With Complex Regional Pain Syndrome (CRPS)
Brief Title: Efficacy of Parecoxib on Patients With CRPS
Status: No longer available | Type: Expanded Access
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Ruhr University of Bochum
Other Study IDs: COX2009; 2009-009433-14 (EudraCT Number)
Record Dates: First submitted 2012-01-31; First posted 2012-02-01 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Causalgia
Keywords: Causalgia; CRPS; complex regional pain syndrome; Dynastat; Parecoxib
MeSH Terms: conditions — Causalgia; Complex Regional Pain Syndromes | interventions — parecoxib

INTERVENTIONS:
Drug: Parecoxib — 90mg Parecoxib i.v. two times a day, two days in a row
  Other Names: Dynastat
Drug: Placebo — NaCl i.v. two times a day, two days in an row
  Other Names: sodium chlorid

SUMMARY:
The complex regional pain syndrom is a weighty disease that often results in a lifelong disability. Mostly this disease appears unilateral after comparatively mundane fractures or operations. In early stages CRPS shows inflammatory processes. These inflammatory components can be seen as edema and vasodilatation. These inflammatory processes lead us to the hypothesis that selective COX-2-inhibitors might help patients with CRPS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with saved diagnosis of CRPS of the upper extremity based on the current used criteria for diagnosis plus a positiv 3-phase-sceletal-scintilgraphy, if they show pathological PPT-values in QST on the ipsilateral site (Z-values > 2 in age- and gender-based Z-transformation of the raw values)• age ≥ 18 years• Existence of an age-based normal creatinin-clearance (calculated with a defined formula)

Exclusion Criteria:

* Important cardiovascular illness for the purpose of heart failure (NYHA II - IV), coronary heart disease (CHD), peripheral artery occlusive disease (PAOD) or unstable hypertension (values constantly over 140/90 mm Hg)

  * Florid kidney disease
  * Cerebral disease
  * Neurological systemic disorder (exception: beginning polyneuropathy with normal values of the PPT on the opposite side)
  * Lesion of the median nerve (ipsi- oder contralateral)
  * Acute bleeding disease
  * Known ulcer of the stomach or duodenum
  * Inflammatory bowel disease
  * Positive anamnesis of a gastrointestinal bleeding in the last 5 years
  * Important hepatic dysfunction (Child- pugh > 9)
  * Hypersensitivity to the agent or to sulfonamides
  * Known allergy to acetylsalicylic acid, nonsteroidal antiinflammatory drugs or other selectiv cyclooxygenase-inhibitors
  * Pregnancy and lactation period
  * Intake of one of the following drugs (current or in the last 3 days)

    * selective-serotonin-reuptake-inhibitor
    * cetoconazole
    * rifampicin
    * phenytoin
    * carbamazepine
    * dexamethasone or other systemic corticoids
    * traditional nonsteroidal antiphlogistics
    * cyclooxygenase-inhibitors
    * immunsupressives
    * TNF-α-inhibitors

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult